CLINICAL TRIAL: NCT01115140
Title: Effect of Metformin With or Without Folate Addiction on Uterine Blood Flow and Trophoblastic Invasion in Pregnant Patients With Polycystic Ovary Syndrome
Brief Title: Metformin and Folate in Pregnant Polycystic Ovary Syndrome(PCOS) Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Department of Obstetrics and Gynecology, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01/2010
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Pregnancy; Polycystic Ovary Syndrome
Keywords: Folate; Metformin; PCOS; Pregnancy; Trophoblastic invasion; Uterine artery velocimetry
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A1 (Active Comparator): metformin plus placebo
  Interventions: Drug: metformin plus placebo
- Group A2 (Experimental): metformin plus folic acid
  Interventions: Drug: Metformin plus folic acid
- Group A3 (Active Comparator): placebo plus folic acid
  Interventions: Drug: placebo plus folic acid
- Group A4 (Placebo Comparator): placebo cp, 2 cps daily
  Interventions: Drug: placebo alone
- Group B (No Intervention): observation

INTERVENTIONS:
Drug: metformin plus placebo — metformin 850 mg cp, 2 cps daily
  Arms: Group A1
Drug: Metformin plus folic acid — metformin 850 mg cp, 2 cps daily plus folic acid 0.4 mg daily
  Arms: Group A2
Drug: placebo plus folic acid — Placebo 1 cp daily plus folic acid 0.4 mg daily
  Arms: Group A3
Drug: placebo alone — placebo cp, 2 cps daily
  Arms: Group A4

SUMMARY:
A more recent prospective nonrandomized placebo-controlled double-blind clinical study demonstrated that metformin exerts a slight but significant deleterious effect on serum homocysteine (Hcy) levels in patients with PCOS, and supplementation with folate is useful to increase the beneficial effect of metformin on the vascular endothelium.

DETAILED DESCRIPTION:
PCOS (cases) and non-PCOS (controls) pregnant women were enrolled. Cases will be randomized in four treatment groups: metformin plus placebo (group A1), metformin plus folic acid (group A2), placebo plus folic acid (group A3), placebo alone (group A4). Controls will not received any treatment (group B). Clinical and biochemical assessment (including serum markers of implantation), Doppler velocimetry of the uterine arteries, and trophoblastic invasion at histological and immunohistochemical evaluation.

Changes in clinical and biochemical data under treatment, pattern of Doppler velocimetry at the uterine arteries, and trophoblastic invasion were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* PCOS

Exclusion Criteria:

* Risk factors for pregnancy complications
* Severe obesity

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Trophoblastic invasion. | two weeks
  Istologic evaluation of trophoblastic ivasion,

SECONDARY OUTCOMES:
Doppler velocimetry measurements of the uterine artery. | two weeks
  Ultrasonographyc assessment of Doppler velocimetry measurements of the uterine artery.

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD, Study Chair — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Catanzaro, Italy